CLINICAL TRIAL: NCT02398916
Title: Effects of Music Listening During Loop Electrosurgical Excision Procedure on Anxiety, Pain, and Satisfaction: a Randomized Controlled Trial
Brief Title: Music Listening to Reduce Pain and Anxiety During LEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kittipat Charoenkwan, MD, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OBG-2557-02665
Record Dates: First submitted 2015-02-27; First posted 2015-03-26 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music (Experimental): * Listening to relaxing music for the entire period starting from waiting period in the surgical waiting area until the end of the LEEP procedure
  * Undergoing LEEP according to the usual protocol
  Interventions: Behavioral: Music listening
- Control (No Intervention): - Undergoing LEEP according to the usual protocol without listening to music

INTERVENTIONS:
Behavioral: Music listening
  Arms: Music

SUMMARY:
Loop electrosurgical excision procedure (LEEP) is the primary diagnostic and therapeutic procedure employed in women with high-grade intraepithelial neoplasia of the cervix. The procedure usually performed in the outpatient setting under local anesthesia. However, it could be associated with significant pain and anxiety.

The aim of this study is to examine the effects of listening to music during the procedure in reducing pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Women with confirmed or suspected high-grade intraepithelial neoplasia of the cervix

Exclusion Criteria:

* Allergy to local anesthetic agent (lidocaine)
* Pregnancy
* Previous major surgical procedures on cervix (conization, LEEP, laser therapy, cryotherapy) or uterus
* Using cardiac pacemaker or history of cardiac arrhythmia
* Neurological disorder affecting perception of pain
* History of lower urinary tract cancer
* Coagulation defects
* History of drug dependence
* Lower genital tract infection
* Apparent invasive cancer of the cervix
* Hearing difficulty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Procedure-related pain, as measured by Visual Analog Scale | During the procedure

SECONDARY OUTCOMES:
Procedure-related anxiety, as measured by Visual Analog Scale | During the procedure
Procedure-related satisfaction, as measured by Visual Analog Scale | During the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kittipat Charoenkwan, MD, Principal Investigator — Faculty of Medicine, Chiang Mai University
Locations (1):
- Department of OB-GYN, Faculty of Medicine, Chiang Mai University, Chiang Mai, Chiang Mai, Thailand